CLINICAL TRIAL: NCT04680455
Title: Potential Benefits of Strength Training for Men Living With Obesity
Brief Title: Strength Training for Men Living With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNew Brunswick
Record Dates: First submitted 2020-12-01; First posted 2020-12-23 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: Physical Activity; Men; Strength Training
MeSH Terms: conditions — Obesity; Motor Activity; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group were asked to exercise three times per week while performing four basic bodyweight exercises in a circuit manner for 12 weeks while supervised online via the Microsoft TEAMs platform. Participants were eased into the program by completing 120 minutes of exercise in week one, 150 minutes in week two, and 180 minutes in the following weeks. Participants were supervised 3X/week for the first four weeks, then 2X/week for the next four weeks and 1X/week for the remaining four weeks. At each session, participants performed the four prescribed exercises (squats, tricep dips, lunges, and push-ups) for 45 seconds each, then switched immediately (15 seconds) to the next exercise followed by one minute of rest at the end of each circuit. Following this exercise program, men living with obesity were able to reach moderate intensity.
  Interventions: Other: Online home-based strength training
- Control (No Intervention): Participants allocated to the control group received an online exercise resource for a 12-week workout plan covering fitness components required to reach both components of the weekly physical activity guidelines on their own. It was recommended that they do a minimum of 150 minutes of moderate to vigorous aerobic activities and two sessions of muscle-strengthening activities using an online program. No supervision was offered and no contact was permitted between the research team and participants from this group.

INTERVENTIONS:
Other: Online home-based strength training — Body weight exercises (i.e., squats, tricep dips, lunges, and push-ups) delivered online through Teams
  Arms: Intervention

SUMMARY:
Emerging evidence suggests that alternative obesity management strategies need to address barriers to engaging with regular physical activity to adopt healthier lifestyles. It is hypothesized that more men living with obesity who are exposed to an online home-based circuit strength training for 12 weeks will be more physically active, 34 weeks after the intervention compared with people who are not exposed to the program.

DETAILED DESCRIPTION:
Sixty men (age ≥ 18 years; body fat % ≥ 25) were randomly assigned to the intervention group (N=30) or the control condition (N=30) for 12 weeks. The intervention group did the online delivered circuit training, three sessions in a week. Adherence to the weekly physical activity guidelines was evaluated 46 weeks after being enrolled in the program using a heart rate tracker and an exercise log. Most variables (anthropometrics, body composition, resting heart rate, blood pressure, lipids profile, glucose) were measured at baseline and after 12, 24, and 46 weeks. Aerobic fitness and comfort with technology were measured at baseline. Perceived benefits/barriers of participation in exercise were captured at baseline and 12 weeks.

More participants in the intervention group adhered to the physical activity guidelines compared to the control group at 46 weeks (intervention 36.8% vs control 5.3%; p=0.021). However, the intervention group did not improve their health outcomes after 12, 24, and 46 weeks. Fewer barriers were reported after 12-week for the intervention group (p=0.02).

ELIGIBILITY:
Inclusion Criteria:

* men
* Body fat% of 25% or more
* Not reaching physical activity guidelines (150 min of moderate to vigorous intensity of aerobic exercises + two sessions of resistance training)
* being able to do weight training

Exclusion Criteria:

- Taking medications that can cause to change in heart rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Representing as men
Enrollment: 60 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Physical activity Level | 48 weeks
  Adherence to the both components of the physical activity guidelines

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline
  Maximum volume of oxygen consumption (Vo2peak)
BMI | 46 weeks
  Anthropometrics
Waist circumference | 46 weeks
  Anthropometrics
Body fat percentage | 46 weeks
  Body composition
Muscle mass | 46 weeks
  Body composition
Metabolic profile | 46 weeks
  High density lipoprotein, low density lipoprotein, triglyceride, resting heart rate, blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keshavarz M, Senechal M, Bouchard DR. Online Circuit Training Increases Adherence to Physical Activity: A Randomized Controlled Trial of Men with Obesity. Med Sci Sports Exerc. 2023 Dec 1;55(12):2308-2315. doi: 10.1249/MSS.0000000000003270. Epub 2023 Aug 2. PMID 37535330

DOCUMENTS (1):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT04680455/Prot_000.pdf